CLINICAL TRIAL: NCT06209008
Title: Efficacy and Safety of Submucosal Intravesical Injection of Platelet-rich Plasma in the Treatment of Interstitial Cystitis/Painful Bladder Syndrome
Brief Title: Submucosal Intravesical Injection of Platelet-rich Plasma in the Treatment of Painful Bladder Syndrome
Acronym: PRP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Younan Ramsis, Lecturer, Ain Shams University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Intravesical injections 001
Record Dates: First submitted 2024-01-02; First posted 2024-01-17 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Painful Bladder Syndrome (PBS); Interstitial Cystitis
Keywords: Platlet Rich Plasma; Intersticial cystitis; Endoscopic Management; Painful bladder syndrome
MeSH Terms: conditions — Cystitis, Interstitial

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intravesical PRP injection (Experimental): Patients will receive 20 submucosal injections of PRP solution, each injection site receives 0.5 mL PRP. The injection needle will be inserted about 1 mm into the at the posterior and lateral walls of the bladder, using a 23 gauge needle and 22 F rigid cystoscope.
  Interventions: Drug: Intravesical injection of Platlet Rich Plasma (PRP)

INTERVENTIONS:
Drug: Intravesical injection of Platlet Rich Plasma (PRP) — Patients will receive 20 submucosal injections of PRP solution, each injection site receives 0.5 mL PRP. The injection needle will be inserted about 1 mm into the at the posterior and lateral walls of the bladder, using a 23 gauge needle and 22 F rigid cystoscope.
  Other Names: PRP intradetrouser injection

SUMMARY:
Interstitial cystitis/painful bladder syndrome (IC/PBS) is characterized by a constellation of bladder symptoms, including urinary frequency, urgency, nocturia, and pelvic pain.

Current intravesical IC/PBS treatment strategies include substances injected submucosally such as botulinum toxin A (BoNTA), or installed intravesically such as bacillus Calmette-Guerin (BCG), resiniferatoxin (RTX), lidocaine, chondroitin sulfate (CS), oxybutynin, and pentosan polysulfate (PPS).

Plasma Rich Protein (PRP) is rich in growth factors, such as platelet-derived growth factor, epidermal growth factor, and transforming growth factor. With the help of these growth factors the defective epithelium can undergo proliferation, differentiation, and wound healing.

DETAILED DESCRIPTION:
A Prospective clinical trial to assess the effectiveness of submucosal intravesical injection of autologous platelet-rich plasma in the treatment of IC/PBS resistant to conventional methods of treatment. It was held in the hospitals of Ain Shams University.

after meeting inclusion and exclusion criteria and attaining the written consent from the patients, they were submitted to intravesical injection of PRP.

All procedures were performed under spinal or general anaesthesia and all patients had received a third generation cephalosporin at the induction of anaesthesia.

Patients received 20 submucosal injections of PRP solution, each injection site receives 0.5 mL PRP. The injection needle was inserted about 1 mm into the at the posterior and lateral walls of the bladder, using a 23 gauge needle and 22 F rigid cystoscope.

After the PRP was injected, a 16 Fr urethral Foley catheter was left for one night to monitor the urine colour and patients were discharged on the next day. Oral antibiotics were prescribed for 3 days.

Patients were followed up in the outpatient clinic after one week with urine culture and then every month after the PRP treatment day. The results of Global Response Assessment (GRA), the O'Leary-Sant score and pain Visual Analogue Scale (VAS) were recorded at baseline, 1, 3 and 6 months after the PRP treatment. The treatment outcome was assessed by the Global Response Assessment (GRA) at 6 months after the PRP injection. The GRA is a seven-point symmetric scale used with the following possible responses: markedly worse (-3), moderately worse (-2), slightly worse (-1), no change (0), slightly improved (+1), moderately improved (+2), and markedly improved (+3). The result was considered as excellent when patients reported improvement in the GRA by >2 or patients became free of bladder pain (VAS = 0). The outcome was considered improved if there is improvement in the GRA by =1 or the pain VAS score reduced by 2. Patients with excellent and improved results were considered as having successful treatment. Otherwise, the treatment was considered to have failed.

Operative time measured in minutes after the induction of anaesthesia.

Complications were recorded associated with the operation including:

* Macroscopic haematuria: detected on the 1st postoperative day.
* Urinary tract infection: detected either by postoperative fever or by positive urine culture collected 1 week postoperatively.

ELIGIBILITY:
Inclusion Criteria:

1. History of symptoms of bladder pain/discomfort related to bladder filling and accompanied by other symptoms such as frequency and urgency.
2. The symptoms are lasting for not less than 6 months.
3. Failed medical treatment in the form of IC/PBS symptoms not relieved by antimicrobials, anticholinergics or antispasmodics after 6 months.

Exclusion Criteria:

1. Pregnancy or lactation.
2. Prior therapy with intravesical treatment.
3. Incomplete medical therapy (Receiving therapy for <3 months with antidepressants, anti-histaminics, hormonal agonists or antagonists).
4. Previous bladder or pelvic surgery or procedure having affected the bladder function.
5. Urodynamic study showing detrusor overactivity.
6. Elevated serum Prostatic Specific Antigen (PSA) level in males
7. Other causes of IC/PBS symptoms including :

   i) Urinary bladder malignancy: bladder masses shown by ultrasonography or malignant cells by urine cytology.

   ii) Indwelling catheters. iii) Infection: urinary tract infection, sexually transmitted disease and vaginitis.

   iv) Chronic bacterial prostatitis. v) Chemical, tuberculous or radiation cystitis. vi) Bladder or lower ureteral calculi by non-contrast computed tomography (CT). vii) Pelvic organ prolapse (POP) by POP-Q assessment system. viii) Bladder outlet obstruction (BOO) diagnosed by urodynamic study.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Global Response Assessment (GRA) at 6 months after the PRP injection. | at 1, 3, 6 months
  The GRA is a seven-point symmetric scale used with the following possible responses: markedly worse (-3), moderately worse (-2), slightly worse (-1), no change (0), slightly improved (+1), moderately improved (+2), and markedly improved (+3). The result was considered as excellent when patients reported improvement in the GRA by >2 and improved if there is improvement in the GRA by =1
Visual Analogue Scale (VAS) | 1, 3, 6 months
  Visual analogue scale is a uni-dimensional measure of pain intensity, used to record patient's pain progression, or compare pain severity between patients with similar conditions. We used a straight horizontal line of fixed length (100 mm), divided into 5 points starting from 0. No pain, 1. Slight discomfort, 2. Bearable pain, 3. Strong Pain and 4. Agonizing unbearable pain.
  The result was considered as excellent when patients reported no bladder pain (VAS = 0).
  The outcome was considered improved if pain VAS score reduced by 2 points on the scale.

SECONDARY OUTCOMES:
Macroscopic hematuria | first postoperative day
  Presence of more than 100 Red blood cells (RBC's) / High power field (HPF) in urine analysis
urinary tract infection | after hospital discharge by 48 hours.
  Doing a nitrate dipstick test that will de done after discharge by 48 hours, if negative indicates that there is no infection. If positive, it is an indication of the presence of UTI, then a culture and senstivity will be ordered and antibiotic prescribed according to it.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed T Hassan, Assisstant Professor, Study Director — AinShams University
Locations (1):
- Demerdash hospital, Faculty of medicine, Ain Shams University, Cairo, Abbassia, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van de Merwe JP, Nordling J, Bouchelouche P, Bouchelouche K, Cervigni M, Daha LK, Elneil S, Fall M, Hohlbrugger G, Irwin P, Mortensen S, van Ophoven A, Osborne JL, Peeker R, Richter B, Riedl C, Sairanen J, Tinzl M, Wyndaele JJ. Diagnostic criteria, classification, and nomenclature for painful bladder syndrome/interstitial cystitis: an ESSIC proposal. Eur Urol. 2008 Jan;53(1):60-7. doi: 10.1016/j.eururo.2007.09.019. Epub 2007 Sep 20. PMID 17900797
- [Background] Pape J, Falconi G, De Mattos Lourenco TR, Doumouchtsis SK, Betschart C. Variations in bladder pain syndrome/interstitial cystitis (IC) definitions, pathogenesis, diagnostics and treatment: a systematic review and evaluation of national and international guidelines. Int Urogynecol J. 2019 Nov;30(11):1795-1805. doi: 10.1007/s00192-019-03970-5. Epub 2019 May 9. PMID 31073635
- [Background] Hanno PM, Erickson D, Moldwin R, Faraday MM; American Urological Association. Diagnosis and treatment of interstitial cystitis/bladder pain syndrome: AUA guideline amendment. J Urol. 2015 May;193(5):1545-53. doi: 10.1016/j.juro.2015.01.086. Epub 2015 Jan 23. PMID 25623737
- [Background] Etulain J. Platelets in wound healing and regenerative medicine. Platelets. 2018 Sep;29(6):556-568. doi: 10.1080/09537104.2018.1430357. Epub 2018 Feb 14. PMID 29442539